CLINICAL TRIAL: NCT02533401
Title: A Multicenter, Single-Arm, Phase II Study to Evaluate the Efficacy and Safety of Rituximab Plus Fludarabine and Cyclophosphamide (FCR) as First-Line Treatment in Patients With B-Cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of Rituximab (MabThera) in Participants With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18429
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-03

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cyclophosphamide; fludarabine; Rituximab

ARMS (1):
- Rituximab + Fludarabine + Cyclophosphamide (Experimental): Participants will receive rituximab (375 milligrams per meter-squared [mg/m^2] intravenously [IV]) on Cycle 1 Day 1, followed by fludarabine (25 mg/m^2 once daily IV) and cyclophosphamide (250 mg/m^2 once daily IV) for Days 2 to 4 of Cycle 1. Then rituximab (500 mg/m^2 IV) will be administered on Day 1 of Cycles 2 to 6, followed by IV fludarabine (25 mg/m^2 once daily IV) and cyclophosphamide (250 mg/m^2 once daily IV) on Days 1 to 3 of Cycles 2 to 6. Each cycle will be 28 days or 4 weeks in length, and the overall duration of treatment will be approximately 6 months.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide will be administered IV at 250 mg/m^2/day on Day 2-4 of Cycle 1 and then on Day 1-3 of Cycles 2 to 6. Each cycle will be 28 days or 4 weeks in length.
Drug: Fludarabine — Fludarabine will be administered IV at 25 mg/m^2/day on Day 2-4 of Cycle 1 and then on Day 1-3 of Cycles 2 to 6. Each cycle will be 28 days or 4 weeks in length.
Drug: Rituximab — Rituximab will be administered IV at 375 mg/m^2 on Day 1 of Cycle 1 and then at 500 mg/m^2 on Day 1 of Cycles 2 to 6. Each cycle will be 28 days or 4 weeks in length.
  Other Names: MabThera/Rituxan

SUMMARY:
This study will evaluate the efficacy and safety of rituximab in combination with chemotherapy (fludarabine and cyclophosphamide) in participants with B-cell CLL.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than or equal to (≥) 18 years of age
* B-cell CLL
* No previous treatment for leukemia

Exclusion Criteria:

* History of other malignancies within 2 years before study entry, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, prostate cancer, or breast cancer
* Comorbid condition requiring long-term (greater than [>] 1 month) systemic corticosteroids during study treatment
* Known infection with hepatitis B or C virus or with human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - La Plata
  - Pilar
  - Rosario
- Caracas, Venezuela

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Participants with CLL received 6 treatment cycles of chemotherapy. Rituximab was administered via intravenous (IV) infusion as 375 milligrams per meter-squared (mg/m^2) on Day 1 of Cycle 1 and as 500 mg/m^2 on Day 1 of Cycles 2 to 6. Fludarabine was given as 25 mg/m^2 daily and cyclophosphamide as 250 mg/m^2 daily, each via IV infusion on Days 2 to 4 during Cycle 1 and on Days 1 to 3 during Cycles 2 to 6. The length of each cycle was 28 days.
Period: Overall Study
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Started | 34
Completed | 23
Not Completed | 11
Not completed — Adverse Event/Intercurrent Disease | 3
Not completed — Death | 5
Not completed — Insufficient Response/Progressed Disease | 1
Not completed — Lost to Follow-up | 1
Not completed — Violation of Selection Criteria | 1

BASELINE CHARACTERISTICS:
Population: All Participants Enrolled: All participants who complied with selection criteria at enrollment.
Groups:
- Rituximab + Fludarabine + Cyclophosphamide: Participants with CLL received 6 treatment cycles of chemotherapy. Rituximab was administered via IV infusion as 375 mg/m^2 on Day 1 of Cycle 1 and as 500 mg/m^2 on Day 1 of Cycles 2 to 6. Fludarabine was given as 25 mg/m^2 daily and cyclophosphamide as 250 mg/m^2 daily, each via IV infusion on Days 2 to 4 during Cycle 1 and on Days 1 to 3 during Cycles 2 to 6. The length of each cycle was 28 days.
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Death or Disease Progression
Description: Treatment response was monitored throughout the study and assessed using standardized criteria. Disease progression was defined as the occurrence of at least one of the following: greater than or equal to (≥) 50 percent (%) increase in the longest diameter of at least two enlarged lymph nodes, increase in spleen and/or liver size by at least 2 centimeters (cm) from Baseline as determined by measurement below the costal margin, or ≥50% increase in the number of circulating lymphocytes. The percentage of participants with death or documented disease progression at any time during the study was calculated.
Time Frame: Up to 5 years (from Baseline until disease progression or death, whichever occurred first)
Population: All Participants Enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
percentage of participants | 24

2. Primary Outcome: Progression-Free Survival (PFS)
Description: Treatment response was monitored throughout the study and assessed using standardized criteria. Disease progression was defined as the occurrence of at least one of the following: ≥50% increase in the longest diameter of at least two enlarged lymph nodes, increase in spleen and/or liver size by at least 2 cm from Baseline as determined by measurement below the costal margin, or ≥50% increase in the number of circulating lymphocytes. PFS was defined as the time from study inclusion until first event of disease progression or death and was estimated using Kaplan-Meier analysis.
Time Frame: Up to 5 years (from Baseline until disease progression or death, whichever occurred first)
Population: All Participants Enrolled.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
months | 47.2 [42.2 to 52.2]

3. Primary Outcome: Percentage of Participants Who Died
Description: Participants were followed for survival throughout the study. The percentage of participants who died of any cause during the study was calculated.
Time Frame: Up to 5 years (from Baseline until death)
Population: All Participants Enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
percentage of participants | 14

4. Primary Outcome: Overall Survival (OS)
Description: Participants were followed for survival throughout the study. OS was defined as the time from study inclusion until death from any cause and was estimated using Kaplan-Meier analysis
Time Frame: Up to 5 years (from Baseline until death)
Population: All Participants Enrolled.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
months | 49.5 [44.8 to 54.2]

5. Primary Outcome: Percentage of Participants With Complete Response (CR), Nodular Partial Response (nPR), or Partial Response (PR)
Description: Treatment response was monitored throughout the study and assessed using standardized criteria. CR was defined as hemoglobin ≥11 grams per deciliter (g/dL), lymphocytes less than (<) 4000 cells per cubic millimeter (cells/mm^3), neutrophils greater than (>) 1500 cells/mm^3, platelets >100,000 cells/mm^3, bone marrow (BM) biopsy with <30% lymphocytes with no lymphocytic infiltrates, no evidence of lymphoid nodules on physical exam, and performance status of 0. PR was defined as >50% decrease in size of enlarged lymph nodes, hepatomegaly, and splenomegaly, with peripheral counts meeting the same criteria as CR or ≥50% improvement from pre-treatment values. Participants with lymphoid nodules on BM biopsy who otherwise met CR criteria were considered nPR. The percentage of participants with each level of best overall response was calculated.
Time Frame: Up to 4 years (assessed every 3 months during 6-month treatment period, every 2 months during 6-month safety follow-up, then every 3 months during 3-year safety follow-up)
Population: All Participants Enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Number analyzed (Participants) | 34
percentage of participants
  CR | 71
  nPR | 9
  PR | 18

ADVERSE EVENTS:
Time Frame: Up to 4 years (assessed every 4 weeks during 6-month treatment period, every 2 months during 6-month safety follow-up, then every 3 months during 3-year safety follow-up
Arm/Group | Rituximab + Fludarabine + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 15/34
Other Adverse Events (participants affected / at risk) | 18/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=34)
Anemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Fever (General disorders) | 3
Infusion related reaction (General disorders) | 1
Febrile neutropenia (Infections and infestations) | 7
Bronchial infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Neoplasm (colon) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures (gallbladder) (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Fludarabine + Cyclophosphamide (N=34)
Anemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 6
Low platelets (Blood and lymphatic system disorders) | 10
Hypogammaglobulinemia (Blood and lymphatic system disorders) | 6
Skin infection (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.